CLINICAL TRIAL: NCT03257449
Title: Effect of Viscous Soluble Fibres on Body Weight Parameters: Review and Meta-analyses
Brief Title: Effect of Viscous Soluble Fibres on Body Weight
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Body Weight Loss Meta
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Overweight and Obesity; T2DM (Type 2 Diabetes Mellitus); General Population
Keywords: Body Weight; Weight loss; BMI; Waist Circumference; Body Fat Percentage; Viscofiber; Viscous Fibres; supplement
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Body Weight; Weight Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Dietary Supplement: Viscous Fibre — Meta-analysis of Randomized Controlled Trials

SUMMARY:
Abstract:

Background: Obesity is a global pandemic affects all age groups and is independent risk factors for most chronic diseases. Dietary intervention is an essential component of obesity management. Dietary fibre supplements have the potential to facilitate weight reduction based on their viscosity. Up to date, the evidence of effects of some fibres on weight is inadequate, and literature provides insufficient information about the effects of the fibre viscosity in weight management.

Objective: Two systematic reviews and meta-analyses of RCTs will be conducted to evaluate the effectiveness of viscous fibres, (agar, alginate, b-glucan from oat and barley, guar gum, glucomannan, pectin, PGX, psyllium), on body weight reduction.

Methods: Only randomised controlled trials are accepted. The trails must have one of the selected fibres as a supplement, and the outcomes must have body weight, BMI, waist circumference, or body fat percentage. Studies shorter than 4 weeks are excluded. Three databases, (Medline, EMBASE, and Cochrane library), were searched through 04/03/2016.

Results: After removing duplicates, 82 studies will be reviewed in full. Significance: This meta-analysis is the first meta-analysis that is based on fibre viscosity, and it will quantify the effect of each fibre in improving weight loss. It will also direct future research in the best direction to further explore this area.

DETAILED DESCRIPTION:
Background: Obesity is a global pandemic and is an independent risk factor for chronic disease. Dietary intervention is an essential component of obesity management. Observational studies show an inverse relationship between dietary fibres and body weight. Therefore, supplements of dietary fibres have the potential to facilitate weight reduction, possibly on the basis of the viscous properties of the fibre. Viscosity is the ability of gel forming that holds water and increase satiety and decreases the amount of intake food. This ability makes dietary fibre supplements considered as appetite suppressants. To date, the evidence of the effect of dietary fibre on weight is inconsistent and controversial and may be dependent on the ability of fibre to induce viscosity. Three previous meta-analyses on Konjac show inconsistency on the effect and its significance. In addition, other meta-analyses on individual viscous fibres show that some viscous fibre does not has an effect on body weight. This is the first meta-analysis that studies the effect of all these fibres together based on their viscosity.

Objective: Two systematic reviews and meta-analyses of RCTs will be conducted to evaluate the effect of viscous and non-viscous fibres on body weight, BMI, waist circumference, and body fat percentage.

Methods: To meet eligibility criteria, the study should be: randomized, controlled, include one of the selected fibres (agar, alginate, b-glucan from oat and barley, guar gum, konjac, pectin, PGX, Psyllium, and xanthan) as a supplement and one of the required outcomes (body weight, BMI, waist circumference or body fat percentage). Studies shorter than 4 weeks in duration will be excluded. Three databases (Medline, EMBASE, and Cochrane Library) were searched. After the search, a title/abstract screening was done to exclude the ineligible articles before extracting data from full eligible studies. Data were extracted using a PROFORMA. Review Manager 5.3 (RevMan) was used to carry out the analysis using generic inverse variance method (GIVM). Change from baseline and standard deviation were utilized in random effect model to get the pooled mean difference effect. Subgroup analyses were done using meta-regression in STATA to explore confounders. GRADE approach was conducted to evaluate the quality of evidence and the strength of recommendations.

Results: Databases were searched through 04/03/2016 and updated on 11/04/2017. Twenty-seven studies were eligible for analyses . The overall effect of viscous fibres on body weight was a significant reduction of -0.38 kg [95%CI: -0.3, -0.13] (P=0.003). BMI, waist circumference and body fat were also significantly reduced: -0.41 kg/m2 [95% CI: -0.61, -0.21](p = 0.0001) -0.78 cm[95%CI: -1.33, -0.24] (p = ) and -1.28 %[95% CI: -2.09, -0.46] (p = ), respectively.

Significance: This study is the first systematic review and meta-analysis that evaluated separately the effect of viscous and non-viscous fibres on weight in the general population. The analysis may help guide diet recommendations for obesity and identify the effect of fibres to direct future research this area.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a randomized controlled clinical trial with either a parallel or cross-over design
2. Must have a treatment period of at least 4 week.
3. Healthy children and adults, overweight and obese individuals or individuals with diabetes were all acceptable
4. Must have one of the selected viscous fibres, (agar, alginate, β-glucan, guar gum, pectin, polyglycoplex(PGX), Psyllium, Xanthan), as a supplemented treatment.
5. Only β-glucan sources from barley or oat were accepted The amount of barley product or barley β-glucan must be reported or measured, or must be computable. β-glucan was considered to be 4.75% in barley, and 3-5% in oat.
6. Must be appropriately controlled.
7. Must measure one of outcomes: body weight, BMI, waist circumference, or Body fat percentage.
8. These Anthropometry measures can be either primary or secondary outcomes.
9. Enough information must be provided to calculate the magnitude of effect, i.e. end of treatment measures and/or change from baseline measures
10. Ad lipitum diet only.

Exclusion Criteria:

1. If the soluble fibre was not one of the selected viscous fibre or a combination.
2. supplement where these fibers could not be isolated each one alone.
3. If the study was insufficiently controlled, i.e. the control was another soluble fibre.
4. If the outcome measures did not include body weight, BMI, waist circumference, or Body fat percentage.
5. If the intervention was a diet with no supplemented fibre.
6. If the study provided insufficient information to calculate a magnitude of effect
7. If the study protocol maintains baseline weight.
8. Secondary information such as reviews, editorials, commentaries, were excluded
9. If the diet is hypo-caloric, energy restricted diet, or metabolically controlled diet.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study includes all population types.
Sampling Method: Probability Sample
Enrollment: 1268 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Body weight chang | in 4 weeks or more
  unit of measure: Kg
BMI change | in 4 weeks or more
  unit of measure: Kg/m2
Waist circumference change | in 4 weeks or more
  unit of measure: Cm
Body fat percentage change | in 4 weeks or more
  unit of measure: %

CONTACTS AND LOCATIONS:
Overall Officials: Nourah Mazhar, MSc (C), Study Director — St.Michael Hospital
Locations (1):
- The Toronto 3D Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jovanovski E, Mazhar N, Komishon A, Khayyat R, Li D, Blanco Mejia S, Khan T, Jenkins AL, Smircic-Duvnjak L, Sievenpiper JL, Vuksan V. Effect of viscous fiber supplementation on obesity indicators in individuals consuming calorie-restricted diets: a systematic review and meta-analysis of randomized controlled trials. Eur J Nutr. 2021 Feb;60(1):101-112. doi: 10.1007/s00394-020-02224-1. Epub 2020 Mar 20. PMID 32198674
- [Derived] Jovanovski E, Mazhar N, Komishon A, Khayyat R, Li D, Blanco Mejia S, Khan T, L Jenkins A, Smircic-Duvnjak L, L Sievenpiper J, Vuksan V. Can dietary viscous fiber affect body weight independently of an energy-restrictive diet? A systematic review and meta-analysis of randomized controlled trials. Am J Clin Nutr. 2020 Feb 1;111(2):471-485. doi: 10.1093/ajcn/nqz292. PMID 31897475